CLINICAL TRIAL: NCT01182207
Title: A Relative Bioavailability Study of 3 mg/0.02 mg Drospirenone/Ethinyl Estradiol Tablets Under Non-Fasting Conditions.
Brief Title: Drospirenone/Ethinyl Estradiol (3 mg/0.02 mg) Tablets Under Non-Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Pharmaceuticals USA (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: R06-0632
Record Dates: First submitted 2010-08-12; First posted 2010-08-16 (Estimated); Results first posted 2010-10-07 (Estimated); Last update posted 2010-12-08 (Estimated); Status verified 2010-11

CONDITIONS: Healthy
Keywords: Bioequivalence; Healthy Subjects
MeSH Terms: interventions — drospirenone; Ethinyl Estradiol; drospirenone and ethinyl estradiol combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Investigational Test Product (Experimental): Drospirenone/Ethinyl Estradiol Tablets, 3 mg/0.02 mg
  Interventions: Drug: Drospirenone/Ethinyl Estradiol (Gianvi®)
- Reference Listed Drug (Active Comparator): YAZ® Tablets, 3 mg/0.02 mg
  Interventions: Drug: YAZ®

INTERVENTIONS:
Drug: Drospirenone/Ethinyl Estradiol (Gianvi®) — 3 mg/0.02 mg Tablets
  Other Names: Gianvi®
  Arms: Investigational Test Product
Drug: YAZ® — 3 mg/0.02 mg Tablets
  Other Names: Drospirenone/Ethinyl Estradiol (generic name)
  Arms: Reference Listed Drug

SUMMARY:
This study was designed to compare the relative bioavailability (rate and extent of absorption) of 3 mg/0.02 mg Drospirenone/Ethinyl Estradiol Tablets with that of YAZ® Tablets (by Berlex, Inc.) following a single, oral dose (2 x 3 mg/0.02 mg tablets) in healthy, adult subjects under non-fasting conditions.

DETAILED DESCRIPTION:
Criteria for Evaluation: FDA Bioequivalence Criteria

Statistical Methods: FDA Bioequivalence Statistical Methods

ELIGIBILITY:
Inclusion Criteria:

* Subjects who were informed of the nature of the study and agreed to read, review, and sign the informed consent document prior to Period I dosing.
* Subjects who completed the screening process within 28 days prior to Period I dosing.
* Subjects who were healthy, adult, menstruating women 18 to 35 years of age, inclusive, at the time of dosing.
* Subjects with a body mass index (BMI) between 19 and 30 kg/m2, inclusive, and weighed at least 110 pounds.
* Subjects who were healthy as documented by the medical history, physical examination, vital sign assessments, 12-lead electrocardiogram, clinical laboratory assessments, and by general observations. The physical examination also included a gynecological exam. If the subject had completed an acceptable Pap smear and gynecological exam in the previous 12 months (prior to study Day 1) and the documentation of acceptable results were provided, both were deferred. Any abnormalities/deviations from thee normal range which were considered clinically relevant by the study physician and investigator were evaluated for individual cases, documented in study files, and agreed upon by the study physician and investigator prior to enrolling a volunteer in the study and for continued enrollment.
* Female subjects who practice an acceptable non-hormonal method of birth control as judged by the investigator(s) at least 14 days prior to Period I dosing, throughout the study, and until 14 days after Period II dosing. The acceptable non-hormonal birth control methods included: double barriers, non-hormone releasing intrauterine device in place for at least 30 days prior to dosing, abstinence throughout the duration of the study, or surgically sterile for at least 6 months prior to Period I dosing.

Exclusion Criteria:

* Volunteers who report receiving any investigational drug within 30 days prior to Period I dosing.
* Volunteers who reported taking any oral contraceptives including estrogen and progestin combined pills and progestin only pills or patch within 28 days prior to Period I dosing, or using injectable contraceptives within 6 months of Period I dosing.
* Volunteers who have ever had progestational hormone implants.
* Volunteers who reported any presence or history of a clinically significant disorder involving the cardiovascular, respiratory, renal, liver, gastrointestinal, immunologic, hematologic, endocrine, or neurologic system(s), or psychiatric or epilepsy disease as determined by the clinical investigator(s).
* Volunteers who reported any presence or history of migraines or severe headaches.
* Volunteers who had a systolic blood pressure lower than 90 or over 140 mmHg, or diastolic blood pressure lower than 45 or over 90 mmHg were excluded from the study.
* Volunteers who had a history of thrombotic disorders, have ever had a cerebrovascular accident, or had transient ischemic attacks.
* Volunteers with a history of breast cancer or undiagnosed breast nodules, active malignancies, or undiagnosed vaginal bleeding.
* Volunteers having other conditions that may be aggravated by fluid retention (as determined by principle investigator).
* Volunteers who had a history of jaundice with previous use of oral contraceptives or any other kinds of hormonal contraceptives.
* Volunteers whose clinical laboratory test values outside the acceptable range and when confirmed on re-examination were deemed to be clinically significant.
* Volunteers who demonstrated a reactive screen for hepatitis B surface antigen, hepatitis C antibody, or HIV antibody.
* Volunteers who reported a history of allergic response(s) to drospirenone/ethinyl estradiol, progestin/estrogens, or related drugs.
* Volunteers who reported the use of any systemic prescription medications in the 14 days prior to Period 1 dosing (with the exception of hormonal contraceptives).
* Volunteers who reported the use of any drug known to induce or inhibit hepatic drug metabolism in the 28 days prior to Period I dosing.
* Volunteers who reported a history of clinically significant allergies including drug allergies.
* Volunteers who reported a clinically significant illness during the 4 weeks prior to Period I dosing (as determined by the clinical investigators).
* Volunteers who reported a history of drug or alcohol addiction or abuse within the past year.
* Volunteers who demonstrated a positive drug abuse screen for the study prior to Period I dose administration.
* Volunteers who used tobacco products in the past 6 months.
* Volunteers who reported donating greater than 150 mL of blood within 30 days prior to Period I dosing. All subjects were advised not to donate blood for 4 weeks after completing the study.
* Volunteers who reported donating plasma within 30 days prior to Period I dosing. All subjects were advised not to donate blood for 4 weeks after completing the study.
* Volunteers who demonstrate a positive pregnancy screen.
* Volunteers who were currently breastfeeding.
* Subjects who had used within the 3 months preceding Period I dosing any vaginally administered estrogen or progestin containing products.
* Any volunteer who engaged in unprotected sexual intercourse during the time interval starting 14 days prior to the first period until 14 days after Period II dosing.
* Volunteers who had a hysterectomy or oophorectomy.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2006-07; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony R Godfrey, Pharm.D., Principal Investigator — PRACS Institute, Ltd.
Locations (1):
- PRACS Institute, Ltd., Fargo, North Dakota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Drospirenone/Ethinyl Estradiol (Test) First: 3 mg/0.02 mg Drospirenone/Ethinyl Estradiol Tablets test product dosed in first period followed by 3 mg/0.02 mg YAZ® Tablets reference product dosed in the second period.
- YAZ® (Reference) First: 3 mg/0.02 mg YAZ® Tablets reference product dosed in first period followed by 3 mg/0.02 mg Drospirenone/Ethinyl Estradiol test product dosed in the second period.
Period: First Intervention
Arm/Group | Drospirenone/Ethinyl Estradiol (Test) First | YAZ® (Reference) First
Started | 18 | 15
Completed | 18 | 14
Not Completed | 0 | 1
Not completed — Positive Hepatitis Results | 0 | 1
Period: Washout of 28 Days
Arm/Group | Drospirenone/Ethinyl Estradiol (Test) First | YAZ® (Reference) First
Started | 18 | 14
Completed | 18 | 14
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Drospirenone/Ethinyl Estradiol (Test) First | YAZ® (Reference) First
Started | 18 | 14
Completed | 17 | 14
Not Completed | 1 | 0
Not completed — Emeses within 1 hour of dosing | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Drospirenone/Ethinyl Estradiol (Test) First | YAZ® (Reference) First | Total
Number analyzed (Participants) | 18 | 15 | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 15 | 33
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 15 | 33
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 17 | 13 | 30
  Hispanic | 0 | 1 | 1
  More than One | 1 | 0 | 1
  American Indian | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 18 | 15 | 33

OUTCOME MEASURES:

1. Primary Outcome: Cmax of Drospirenone(Maximum Observed Concentration of Drug Substance in Plasma)
Description: Bioequivalence based on Drospirenone Cmax.
Time Frame: Blood samples collected over a 120 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Drospirenone/Ethinyl Estradiol (Test): 3 mg/0.02 mg Drospirenone/Ethinyl Estradiol Tablets test product dosed in either period.
- YAZ® (Reference): 3 mg/0.02 mg YAZ® Tablets reference product dosed in either period.
Arm/Group | Drospirenone/Ethinyl Estradiol (Test) | YAZ® (Reference)
Number analyzed (Participants) | 31 | 31
ng/mL | 52.77 (15.77) | 53.65 (13.82)
Statistical Analysis 1: Comparison: Drospirenone/Ethinyl Estradiol (Test) vs YAZ® (Reference); Test type: Non-Inferiority or Equivalence — ANOVA is to be used to identify the source contributions by factors including subjects, period, formulation and potential interactions. The geometric mean ratio together with the ANOVA residual mean error term are used to identify the statistical basis for the 90% confidence interval for the ratio of the population means (Test [T]/Reference[R]) of the identified metrics (e.g. AUC, Cmax); Ratio of the T/R geometric mean x 100 = 96.74, 90% CI 2-sided [86.82 to 107.79] — Bioequivalence is established if the 90% confidence interval for the ln-transformed geometric mean between the reference (R) and test (T) product fall within the interval of 80-125%

2. Primary Outcome: AUC0-t of Drospirenone(Area Under the Concentration-time Curve From Time Zero to Time of Last Measurable Concentration)
Description: Bioequivalence based on Drospirenone AUC0-t.
Time Frame: Blood samples collected over a 120 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Drospirenone/Ethinyl Estradiol (Test) | YAZ® (Reference)
Number analyzed (Participants) | 31 | 31
ng*h/mL | 889.67 (187.51) | 867.10 (207.11)
Statistical Analysis 1: Comparison: Drospirenone/Ethinyl Estradiol (Test) vs YAZ® (Reference); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 103.16, 90% CI 2-sided [101.10 to 105.27] — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: AUC0-inf of Drospirenone(Area Under the Concentration-time Curve From Time Zero to Infinity)
Description: Bioequivalence based on Drospirenone AUC0-inf.
Time Frame: Blood samples collected over a 120 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Drospirenone/Ethinyl Estradiol (Test) | YAZ® (Reference)
Number analyzed (Participants) | 31 | 31
ng*h/mL | 951.18 (226.13) | 930.38 (236.38)
Statistical Analysis 1: Comparison: Drospirenone/Ethinyl Estradiol (Test) vs YAZ® (Reference); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 102.72, 90% CI 2-sided [100.67 to 104.80] — [estimate comment as in outcome 1, analysis 1]

4. Primary Outcome: Cmax of Ethinyl Estradiol(Maximum Observed Concentration of Drug Substance in Plasma)
Description: Bioequivalence based on Ethinyl Estradiol Cmax.
Time Frame: Blood samples collected over a 72 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Drospirenone/Ethinyl Estradiol (Test) | YAZ® (Reference)
Number analyzed (Participants) | 31 | 31
pg/mL | 87.95 (29.22) | 91.23 (36.79)
Statistical Analysis 1: Comparison: Drospirenone/Ethinyl Estradiol (Test) vs YAZ® (Reference); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 97.60, 90% CI 2-sided [89.45 to 106.50] — [estimate comment as in outcome 1, analysis 1]

5. Primary Outcome: AUC0-t of Ethinyl Estradiol(Area Under the Concentration-time Curve From Time Zero to Time of Last Measurable Concentration)
Description: Bioequivalence based on Ethinyl Estradiol AUC0-t.
Time Frame: Blood samples collected over a 72 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: pg*h/mL
Arm/Group | Drospirenone/Ethinyl Estradiol (Test) | YAZ® (Reference)
Number analyzed (Participants) | 31 | 31
pg*h/mL | 1066.24 (372.97) | 1079.54 (344.21)
Statistical Analysis 1: Comparison: Drospirenone/Ethinyl Estradiol (Test) vs YAZ® (Reference); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 98.88, 90% CI 2-sided [95.62 to 102.25] — [estimate comment as in outcome 1, analysis 1]

6. Primary Outcome: AUC0-inf of Ethinyl Estradiol(Area Under the Concentration-time Curve From Time Zero to Infinity)
Description: Bioequivalence based on Ethinyl Estradiol AUC0-inf.
Time Frame: Blood samples collected over a 72 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: pg*h/mL
Arm/Group | Drospirenone/Ethinyl Estradiol (Test) | YAZ® (Reference)
Number analyzed (Participants) | 31 | 31
pg*h/mL | 1155.69 (394.56) | 1175.76 (358.58)
Statistical Analysis 1: Comparison: Drospirenone/Ethinyl Estradiol (Test) vs YAZ® (Reference); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 98.20, 90% CI 2-sided [95.36 to 101.12] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over the course of the study, which was approximately 6 weeks in duration.
Description: Volunteers were monitored throughout the study for any adverse experiences. AEs were collected through both solicited and unsolicited methods. The volunteers were encouraged to report signs, symptoms, and any changes in health to the clinic staff.
Arm/Group | Drospirenone/Ethinyl Estradiol (Test) | YAZ® (Reference)
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/33
Other Adverse Events (participants affected / at risk) | 21/33 | 11/33
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Drospirenone/Ethinyl Estradiol (Test) (N=33) | YAZ® (Reference) (N=33)
Nausea (General disorders) | 6 (7) | 4 (4)
Dysmenorrhoea (General disorders) | 4 (4) | 2 (2)
Metrorrhagia (General disorders) | 2 (2) | 3 (3)
Abdominal Pain (General disorders) | 3 (4) | 4 (4)
Vomitting (General disorders) | 3 (6) | 2 (2)
Pharynogolaryngeal Pain (General disorders) | 3 (3) | 0 (0)
Headache (General disorders) | 8 (9) | 3 (3)
Sinus Headache (General disorders) | 2 (2) | 0 (0)
Menstrual Disorder (General disorders) | 1 (1) | 2 (2)
Stomach Discomfort (General disorders) | 2 (2) | 0 (0)
Dizziness (General disorders) | 2 (2) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Principal Investigator is not permitted to discuss or publish trial results.